CLINICAL TRIAL: NCT01596205
Title: The Efficacy of Robot Assisted Group Cognitive Training in Elderly Adults Without Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2011-04-080
Record Dates: First submitted 2012-05-09; First posted 2012-05-10 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Age-Related Cognitive Decline
Keywords: cognitive therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Robot intervention (Experimental): Participants were given baseline assessments and randomly assigned into 3 groups; 24 with robot assisted cognitive training group (Robot intervention group), 24 with experienced behavioral therapist group (Conventional intervention group), and 37 without cognitive training (Control group).It was explained that there was a waiting list, therefore, participants in control group had an opportunity to participate in cognitive training program after a delay of 12 weeks for the intervention.
  Interventions: Behavioral: Robot assisted cognitive training
- Conventional intervention (Active Comparator): conventional cognitive training group - pen and pencil with experienced behavioral therapists
  Interventions: Behavioral: Conventional cognitive training group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Robot assisted cognitive training — We developed total 17 software programs for cognitive training with robot which were intended to develop for improvement of following cognitive function;5 programs for memory, 2 for language , 1 for reasoning, 3 for working memory or speed of processing, 2 for calculation and 4 for visuospatial function.
  Arms: Robot intervention
Behavioral: Conventional cognitive training group — Experienced behavioral therapists who had been clinical neuropsychologists for 2 years instructed the participants in cognitive training. Thearpists were familiarized with manuals for cognitive training before study inception, and were instructed to adhere to the manual but were allowed to distribute time flexibly among the programs in the same cognitive domain.
  In all sessions of conventional intervention group, the behavioral therapists showed several questions or instructions on the screen and then the participants answered to the questions with verbal or written words using paper and pencil.
  Arms: Conventional intervention

SUMMARY:
Previous studies about cognitive intervention targeting older adults revealed that cognitive training had effects on the improvement of cognitive function.However, researches are rare that investigated direct changes of brain structures after cognitive training.

The advanced scientific technique allowed us to develop service robots designed to assist human work, which can be important with an increase in the aging population and high costs of elderly care. In this regard, the investigators considered robots for elderly's cognitive training and developed 17 cognitive programs in collaboration with Center for Intelligent Robotics at Korea Institute of Science and Technology.

The purposes of this study were to demonstrate the effects of the investigators newly developed robot assisted group cognitive training programs on the brain in older adults and to identify whether they can help to improve cognitive function or mood in the elderly compared to the conventional cognitive training or control group that were not involved in any cognitive training.

DETAILED DESCRIPTION:
Primary outcome The primary outcome of this study was the change in cortical thickness between the baseline and the post-intervention assessment.

Secondary outcomes Change in the brain functional network from the baseline to the postintervention assessment was also assessed as a secondary outcome ascertained by the analysis of resting state fMRI, which has been used to show correlated spontaneous activity within cortical and subcortical regions that are functionally related.

Further secondary outcomes were changes between the baseline and the post-intervention assessment on cognitive function measured by validated neuropsychological tests such as SNSB and CANTAB on participants' depressive and anxiety symptoms scored by Geriatric Depression Scale and Geriatric Anxiety Inventory respectively, on self reported memory problems measured by Korean Dementia Screenng Questionnaire, Multifactorial Memory Questionnaire and Prospective and Retrospective Memory Questionnaire, on functions of daily living acitivity measured by Bayer ADL, on quality of life measuared by WHOQOL-bref.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling volunteers aged 60 years or older
* without dementia
* MMSE=26 or above

Exclusion Criteria:

* if they had known dementia or significant cognitive impairment accompanied by dysfunction of daily living activities;
* had 6 years of education or under;
* were illiterate
* were unavailable during the testing and intervention periods of the study;
* had severe losses in vision or hearing; had major neurological or psychiatric illness history including any history of stroke, transient ischemic attack or traumatic brain injury;
* had a medication history which might affect on cognitive function such as acetylcholinesterase inhibitor or memantine
* had medical problems such as thyroid, liver and renal disease;
* had a significan structural abnormalities on their baseline brain MRI.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2011-06; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
the change in cortical thickness between the baseline and the post-intervention assessment. | between the baseline and the post-intervention assessment (12 week training)
  The primary outcome of this study was the change in cortical thickness between the baseline and the post-intervention assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Duk L. Na, MD,PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim GH, Jeon S, Im K, Kwon H, Lee BH, Kim GY, Jeong H, Han NE, Seo SW, Cho H, Noh Y, Park SE, Kim H, Hwang JW, Yoon CW, Kim HJ, Ye BS, Chin JH, Kim JH, Suh MK, Lee JM, Kim ST, Choi MT, Kim MS, Heilman KM, Jeong JH, Na DL. Structural brain changes after traditional and robot-assisted multi-domain cognitive training in community-dwelling healthy elderly. PLoS One. 2015 Apr 21;10(4):e0123251. doi: 10.1371/journal.pone.0123251. eCollection 2015. PMID 25898367